CLINICAL TRIAL: NCT04076267
Title: Psychometric Validation of the French Version of the Modified Edmonton Symptom Assessment Scale: The ESAS12-F.
Brief Title: Psychometric Validation of the ESAS12-F
Acronym: ESAS12-F
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ESAS12-F
Record Dates: First submitted 2019-08-07; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cancer
  Interventions: Other: Tool assessing symptoms validation

INTERVENTIONS:
Other: Tool assessing symptoms validation — Comparison between 2 tools evaluating the symptoms of patients with advanced cancer: the ESAS12-F and the EORTC QLQ C30 to assess if the ESAS12-F well evaluates the symptoms and if it is easy to complete. The objective is to validate the ESAS12-F, which is easier and shorter than the well validated EORTC QLQ C30

SUMMARY:
Assessing symptoms of patients with cancer should be a priority for the physicians to improve their quality of life. The Edmonton Symptom Assessment Scale (ESAS) is a common tool, easy to complete and to analyse. Originally, it has been validated in English with 9 common symptoms. But a new version with 12 commons symptoms and some explanations has been created. This modified version has been translated in French, and the transcultural validation has been done. But the psychometreic validation has not been validated yet.

The primary objective is to validate the psychometric properties of this new version in French.

To validate the tool, we will compare the ESAS12-F to the European Organization for research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) which assesses common symptoms for patients with cancer, which is validated in French, but which is longer and more difficult to complete and to analyse. the patient will complete the ESAS 12-F and the EORTC QLQ-C30 at day 1, then the ESAS12-F at day 2, and the ESAS12-F and the EORTC QLQ-C30 at day 7.

ELIGIBILITY:
Inclusion Criteria:

* more than 18YO
* with advanced cancer
* followed but the palliative care team of the Centre Hospitalier Lyon Sud
* without any cognitive impairment
* can read and speak French

Exclusion Criteria:

* cognitive impairment
* bad performance status
* cannot read or speak French
* no advanced cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than18 YO with advanced cancer, followed by the palliative care team, without any cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
validation of the psychometric properties of the French version of the modified Edmonton Symptom Assessment Scale, the ESAS12-F: construct validity | day 1
  The validation of the French version of the modified ESAS scale will be made by assessing the following metrological properties: validity (criterion validity and construct validity) :
  Criterion validity will be established against the EORTC QLQ-C30 scale using correlation coefficient for each item. It will be assessed at Day 1 and Day 7. Construct validity will be assessed by a principal component analysis (PCA) an exploratory factor analysis (EFA) and then a confirmatory analysis (CFA) on an independent sample.
validation of the psychometric properties of the French version of the modified Edmonton Symptom Assessment Scale, the ESAS12-F: construct validity | day 2
  The validation of the French version of the modified ESAS scale will be made by assessing the following metrological properties: validity (criterion validity and construct validity) :
  Criterion validity will be established against the EORTC QLQ-C30 scale using correlation coefficient for each item. It will be assessed at Day 1 and Day 7. Construct validity will be assessed by a principal component analysis (PCA) an exploratory factor analysis (EFA) and then a confirmatory analysis (CFA) on an independent sample.
validation of the psychometric properties of the French version of the modified Edmonton Symptom Assessment Scale, the ESAS12-F: construct validity | day 7
  The validation of the French version of the modified ESAS scale will be made by assessing the following metrological properties: validity (criterion validity and construct validity) :
  Criterion validity will be established against the EORTC QLQ-C30 scale using correlation coefficient for each item. It will be assessed at Day 1 and Day 7. Construct validity will be assessed by a principal component analysis (PCA) an exploratory factor analysis (EFA) and then a confirmatory analysis (CFA) on an independent sample.
validation of the psychometric properties of the French version of the modified Edmonton Symptom Assessment Scale, the ESAS12-F: test-retest reliability | day 2
  The validation of the French version of the modified ESAS scale will be made by assessing the following metrological properties: reliability (internal consistency and test-retest reliability) :
  Internal consistency will be checked using Cronbach's alpha coefficient or a more adequate coefficient whenever the former is not applicable. Test-retest reliability will be checked using the intra-class correlation coefficient. It will be assessed at Day 2 and Day 7.
validation of the psychometric properties of the French version of the modified Edmonton Symptom Assessment Scale, the ESAS12-F: test-retest reliability | day 7
  The validation of the French version of the modified ESAS scale will be made by assessing the following metrological properties: reliability (internal consistency and test-retest reliability) :
  Internal consistency will be checked using Cronbach's alpha coefficient or a more adequate coefficient whenever the former is not applicable. Test-retest reliability will be checked using the intra-class correlation coefficient. It will be assessed at Day 2 and Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Colombe TRICOU, MD, Study Director — Hospices Civils de Lyon, Université Claude Bernard Lyon 1
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France